CLINICAL TRIAL: NCT01333241
Title: Community-Based Lifestyle Promotion With Latino Women
Brief Title: Healthy Lifestyle Behavior Intervention for Latino Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Deborah Koniak-Griffin, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: G090405102; R01HL086931-A1 (Other Grant/Funding Number: NHLBI (ARRA grant)); R01HL086931 (NIH)
Record Dates: First submitted 2011-04-06; First posted 2011-04-11 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Cardiovascular Diseases
Keywords: Hispanic/Latina Americans; Cardiovascular diseases; Obesity; Intervention
MeSH Terms: conditions — Cardiovascular Diseases; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle behavior intervention group (Experimental): The 6-month lifestyle behavior intervention includes group education and individual teaching and coaching.
  Interventions: Behavioral: Lifestyle behavior interventon grop
- Control group (Sham Comparator): Disaster Preparedness/Home Safety group education and teaching
  Interventions: Other: Placebo Comparator: Control group

INTERVENTIONS:
Behavioral: Lifestyle behavior interventon grop
  Arms: Lifestyle behavior intervention group
Other: Placebo Comparator: Control group
  Other Names: Disaster Preparedness/Home Safety
  Arms: Control group

SUMMARY:
The overall goal of this randomized controlled trial is to evaluate the effects of a community-based lifestyle behavior intervention (LSBI) that is designed to improve dietary habits and physical activity (PA), and reduce weight of Latino women who are predominantly Spanish-speaking immigrants. It is hypothesized that middle-aged overweight/obese Latinas participating in a LSBI conducted by lay health advisors will demonstrate improved dietary habits, increased physical activity and a decrease in BMI compared to those in a control condition, Women in the LSBI also are expected to demonstrate improvements in selected physiologic outcomes (waist circumference, blood pressure [BP], measures of cholesterol and blood sugar).

DETAILED DESCRIPTION:
Overweight/obesity and physical inactivity are two significant predictors of illness and death from cardiovascular (heart) disease (CVD) in Latina adults. These risk factors may be reduced or eliminated through prevention efforts that focus on heart-healthy diets, weight reduction, and PA. The purpose of this study is to compare the effects of a 6-month community-based lifestyle behavior intervention (LSBI) conducted by lay health advisors and a control condition (disaster preparedness and home safety program) on lifestyle behaviors -dietary habits and physical activity(primary outcome) and selected physiologic outcomes (secondary outcomes) i.e., BMI, waist circumference, blood pressure, measures of cholesterol,and fasting blood sugar of Latinas who are overweight/obese. The LSBI includes group education (8 classes) and individual teaching and coaching (8 contacts by home visits and telephone calls) delivered over a 6-month period. Acceptability and feasibility of the intervention is evaluated through examination of women's retention rates and participation in classes and home visits.

ELIGIBILITY:
Inclusion Criteria:

* Latina
* 35 to 64 years of age
* body mass index (BMI) >25
* fluent in either Spanish or English.

Exclusion Criteria:

* pregnant or planning to get pregnant in next year
* history of myocardial infarction or stroke
* currently under treatment for cancer
* orthopedic or joint problems that would prohibit participation in physical activity
* insulin-dependent diabetes

Ages: 35 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 223 (Actual)
Dates: Start 2009-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change in Body mass index (BMI) | Baseline, 6 and 9 month follow-up.

SECONDARY OUTCOMES:
Change in Physical Activity | Baseline, 6 and 9 month follow-up
  Physical activity as determined by accelerometer readings,
Change in Physiologic measures | Baseline, 6 and 9 month follow-up.
  Blood pressure, cholesterol (total, HDL, LDL, and triglycerides), fasting blood sugar, and waist circumference.
Change in Lifestyle behaviors | Baseline, 6 and 9 month follow-up.
  Self-reported eating and physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Koniak-Griffin, RNC, EdD, Principal Investigator — UCLA School of Nursing
Locations (1):
- UCLA School of Nursing, Los Angeles, California, United States

REFERENCES:
- [Background] Koniak-Griffin, D., Brecht, M. L., Takayanagi, S., Villegas, J., Melendrez, M., & Balcázar, H. (2014). A community health worker-led lifestyle behavior intervention for Latina (Hispanic) women: Feasibility and outcomes of a randomized controlled trial. International journal of nursing studies. Koniak-Griffin, D., & Brecht, M.-L. (2014, July 30). Awareness of Cardiovascular Disease and Preventive Behaviors Among Overweight Immigrant Latinas. Journal of Cardiovascular Nursing [Epub ahead of print] Koniak-Griffin, D., Brecht, M. L., Takayanagi, S., Villegas, J., & Melendrez, M. (2013). Physical Activity and Cardiometabolic Characteristics in Overweight Latina Women. Journal of Immigrant and Minority Health, 1-9.
- [Derived] Koniak-Griffin D, Brecht ML, Takayanagi S, Villegas J, Melendrez M, Balcazar H. A community health worker-led lifestyle behavior intervention for Latina (Hispanic) women: feasibility and outcomes of a randomized controlled trial. Int J Nurs Stud. 2015 Jan;52(1):75-87. doi: 10.1016/j.ijnurstu.2014.09.005. Epub 2014 Sep 22. PMID 25307195
- [Derived] Koniak-Griffin D, Brecht ML, Takayanagi S, Villegas J, Melendrez M. Physical activity and cardiometabolic characteristics in overweight Latina women. J Immigr Minor Health. 2014 Oct;16(5):856-64. doi: 10.1007/s10903-013-9782-z. PMID 23355122